CLINICAL TRIAL: NCT04205591
Title: Split Bone Block Technique: Clinical and Radiographic Study Between Autologous and Porcine Xenogeneic Cortical Plates. Randomized Clinical Trial
Brief Title: Comparative Study Between Porcine and Autologous Cortical Plates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Jesús Torres García Denche, Associate Professor, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P-15/567
Record Dates: First submitted 2019-12-15; First posted 2019-12-19 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Bone Regeneration
Keywords: split bone block; RCT

STUDY DESIGN:
Intervention Model Description: 16 patients referred for implant placement and with insufficient bucco-lingual (BL) alveolar bone width (<4 mm) were included in the study.. Patients included in the clinical trial were randomly allocated by a blinded assistant in two groups: in the autogenous cortical plate group (ACP), and xenogeneic cortical plate group (XCP).
Who Masked: Participant, Investigator
Masking Description: Bone augmentation procedures using autogenous cortical plates or xenograft cortical plates were carried on, both using autogenous bone chips to fill the resulting gap. Patients included in this clinical trial were randomly allocated by a blinded assistant in two groups: Autogenous Cortical Plates (ACP) and Xenograft Cortical Plates (XCP). Random allocation of participants to intervention groups was performed using a computerized random number generated by the GraphPad- QuickCalc software (GraphPad Soft- ware Inc., La Jolla, CA) As a result, 9 patients were randomly assigned to de ACP group and 9 to the XCP group. All surgeries were performed by the same oral surgeon (JT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autologous cortical plate (Active Comparator): Thin autologous cortical plates that allow to made a rigid and resistant framework that will be filled with autogenous bone chips bone
  Interventions: Procedure: split bone block technique
- Porcine cortical plate (Experimental): Thin porcine cortical platesthat allow to made a rigid and resistant framework that will be filled with autogenous bone chips bone
  Interventions: Procedure: split bone block technique

INTERVENTIONS:
Procedure: split bone block technique — A graft surgery using autogenous bone chips surrounded by a rigid framework made over the atrophic sites of the mandible and maxilla to obtain bone augmentation to support dental implants

SUMMARY:
The aim of this study is to evaluate the outcome of three-dimensional bone regeneration procedures using thin cortical porcine xenograft plates in combination with autogenous bone chips compared with thin autogenous cortical plates and autogenous bone chips.

DETAILED DESCRIPTION:
Materials and methods: 16 patients referred for implant placement and with insufficient bucco-lingual (BL) alveolar bone width (<4 mm) were included in the study. Patients received autogenous cortical plates (ACP) of either porcine xenogeneic (XCP). The aforementioned groups were compared in regards to bone augmentation using General Estimating Equations (GEE) and logistic regression. Demographic data, trabecular bone density, graft site, postoperative pain, and time consuming were also analyzed

ELIGIBILITY:
Inclusion Criteria:

- Patients were enrolled in the study on the basis of having insufficient bone height (<6mm), width (<3mm) or both, in either maxilla or mandible

Exclusion Criteria:

Patients with severe systemic disease (American Society of Anesthesiology III or IV) were excluded from the study.

In addition, patients who were pregnant, or patients with diseases affecting bone, such as:Paget's disease, osteomalacia, diabetes, vitamin D deficiency, alcoholism, hyperthyroidism cancer or osteoporosis as well as those on medications that might affect bone metabolism, such as bisphosphonates, corticosteroids or antiepileptic medicaments were also excluded from the study.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-05-10 (Actual); Primary Completion 2017-09-08 (Actual); Study Completion 2019-09-13 (Actual)

PRIMARY OUTCOMES:
Volume of bone augmentation | 4 months
  Volume of bone augmentation of the surgical sites was measured in the postoperative parasagittal CT scans using a region of interest (ROI) containing the entire bone box regenerated area using the closed polygon tool of the OsiriX software. This measurements have been done in mm3

SECONDARY OUTCOMES:
Postoperative pain | 4 months
  The amount of pain was classified into three categories: heavy pain, with the patient taking more than eight painkillers (ibuprofen 400); moderate pain, when the patient took four to eight painkillers; or little pain, when the patient needed fewer than four painkillers.
Bone box time consuming | Minutes
  In the control group this was measured from the moment the osteotomy incision began with the MicroSaw until the bone block was completely removed, splitting cortical plates and fixation to the buccal and lingual/palatal side of the bone defect using osteosynthesis screws after it is filled with the bone chips harvested previously. In experimental group the time was measured from the open of porcine cortical plate envelope until the bone box was completely filled and sealed.

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Torres, Associate, Principal Investigator — Universidad Complutense de Madrid

IPD SHARING:
Plan to Share IPD: No